CLINICAL TRIAL: NCT05891080
Title: Neoadjuvant Therapy With Toripalimab and JS004 Combined With Platinum-based Doublet Chemotherapy for Resectable or Potentially Resectable Stage III Non-small Cell Lung Cancer: A Randomised Controlled, Open-label, Phase 2 Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-014
Record Dates: First submitted 2023-05-22; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Stage III Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab; Pemetrexed; 130-nm albumin-bound paclitaxel; Carboplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Safety run-in arm (Experimental): In this arm, 6 patients with resectable or potentially resectable stage III non-small cell lung cancer will receive 4 circles of neoadjuvant toripalimab and JS004 combined with platinum-based doublet chemotherapy and those resectable after neoadjuvant therapy will be treated with surgery.
  Interventions: Drug: Toripalimab; Drug: JS004; Drug: Pemetrexed; Drug: Nab-paclitaxel; Drug: Carboplatin; Procedure: Surgery
- JS004 arm (Experimental): Patients with resectable or potentially resectable stage III non-small cell lung cancer will be randomized into this arm (59 patients) and receive 4 circles of neoadjuvant toripalimab and JS004 combined with platinum-based doublet chemotherapy and those resectable after neoadjuvant therapy will be treated with surgery.
  Interventions: Drug: Toripalimab; Drug: JS004; Drug: Pemetrexed; Drug: Nab-paclitaxel; Drug: Carboplatin; Procedure: Surgery
- Control arm (Active Comparator): Patients with resectable or potentially resectable stage III non-small cell lung cancer will be randomized into this arm (59 patients) and receive 4 circles of neoadjuvant toripalimab combined with platinum-based doublet chemotherapy and those resectable after neoadjuvant therapy will be treated with surgery.
  Interventions: Drug: Toripalimab; Drug: Pemetrexed; Drug: Nab-paclitaxel; Drug: Carboplatin; Procedure: Surgery

INTERVENTIONS:
Drug: Toripalimab — Specified dose on specified days.
Drug: JS004 — Specified dose on specified days.
  Arms: JS004 arm; Safety run-in arm
Drug: Pemetrexed — Specified dose on specified days.
Drug: Nab-paclitaxel — Specified dose on specified days.
Drug: Carboplatin — Specified dose on specified days.
Procedure: Surgery — Patients with resectable tumor after neoadjuvant therapy will be treated with surgery.

SUMMARY:
For stage III non-small cell lung cancer (NSCLC), neoadjuvant chemotherapy plus PD-1 antibody is recommended. However, most patients could not achieve complete pathological response (CPR). New immunotherapeutic strategy is needed to achieve higher CPR rate. JS004 is a new antibody targeting B and T lymphocyte attenuator (BTLA) which restrains the function of immune cells and leads to immune escape of tumor cells. The combination of PD-1 antibody and BTLA antibody has shown good therapeutic effect in solid tumors. This trial aims to investigate the efficacy and safety of the therapeutic regimen of toripalimab and JS004 plus chemotherapy in stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form.
2. Aged 18 ≥ years.
3. Histological or cytological diagnosis of NSCLC by needle biopsy, and stage IIIB-IIIC confirmed by imageological examinations (CT, PET-CT or EBUS).
4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
5. Life expectancy is at least 12 weeks.
6. At least 1 measurable lesion according to RECIST 1.1.
7. Patients with good function of other main organs (liver, kidney, blood system, etc.)
8. Patients with lung function can tolerate surgery;
9. Without systematic metastasis (including M1a, M1b and M1c);
10. Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of toripalimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
11. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 days after chemotherapy or the last dose of toripalimab (whichever is later).

Exclusion Criteria:

1. Participants who have received any systemic anti-cancer treatment for thymic epithelial tumor, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment;
2. Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
3. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment;
4. Participants who are allergic to the test drug or any auxiliary materials;
5. Participants with Interstitial lung disease currently;
6. Participants with active hepatitis B, hepatitis C or HIV;
7. Pregnant or lactating women;
8. Participants suffering from nervous system diseases or mental diseases that cannot cooperate;
9. Participated in another therapeutic clinical study;
10. Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (PCR) rate | Up to 30 months
  PCR rate is defined as the proportion of participants who have achieved pathologic complete response (on routine hematoxylin and eosin staining, no tumor cell can be found in tumor bed or lymph node) in all participants.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 30 months
  ORR is defined according to the RECIST v1.1 criteria.
Major pathologic response (MPR) rate | Up to 30 months
  MPR rate is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants.
Treatment-related adverse event (TRAE) | Up to 30 months
  TRAE is defined and classified according to NCI-CTCAE v5.0 in all participants.
Rate of conversion from potentially resectable to resectable | Up to 30 months
  Rate of conversion from potentially resectable to resectable is defined as the proportion of participants with potentially resectable tumor conversed into resectable tumor in all participants with potentially resectable tumor.
R0 resection rate | Up to 30 months
  R0 resection rate is defined as the proportion of participants who have achieved R0 resection (complete resection with no residual tumor cell in the resection margin) in all participants.
Event-free survival (EFS) | up to 60 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Overall survival (OS) | up to 60 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
EORTC-QLQ-C30 scale | up to 5 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30, Version 3). EORTC's QLQ-C30 (V3.0) is a core scale for lung cancer patients, with a total of 30 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.
EORTC-QLQ-L13 scale | up to 5 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-LC13). EORTC's QLQ-LC13 is a core scale for lung cancer patients, with a total of 13 items. The items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Zhang, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.